CLINICAL TRIAL: NCT03013036
Title: Ultrasonographic Thyrohyoid Distance Measurement for Prediction of Difficult Intubation and Ultrasonographic Prediction of Pediatric Endotracheal Tube Size
Brief Title: Ultrasonography for Prediction of Difficult Intubation and Prediction of Endotracheal Tube Size
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Elif Aybike Ozmumcu, Medical Doctor, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0964
Record Dates: First submitted 2016-12-27; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Intubation; Difficult or Failed
MeSH Terms: interventions — Ultrasonography; Sevoflurane; Propofol; Fentanyl; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (Other): Patients between 1 and 2 years
  Interventions: Device: Ultrasonography; Drug: Sevoflurane; Drug: intravenous midazolam; Drug: fentanyl and rocuronium
- Group II (Other): patients between 3 and 5 years
  Interventions: Device: Ultrasonography; Drug: Sevoflurane; Drug: Propofol; Drug: fentanyl and rocuronium
- Group III (Other): patients between 6 and 8 years
  Interventions: Device: Ultrasonography; Drug: Sevoflurane; Drug: intravenous midazolam; Drug: fentanyl and rocuronium

INTERVENTIONS:
Device: Ultrasonography
Drug: Sevoflurane
Drug: intravenous midazolam
  Arms: Group I; Group III
Drug: Propofol
  Arms: Group II
Drug: fentanyl and rocuronium

SUMMARY:
Aim of our study is to evaluate the predictive value of ultrasonographic (USG) measurement of thyrohyoid distance for difficult intubation and determination of optimal endotracheal tube size by using USG in pediatric patients undergoing elective surgery.

DETAILED DESCRIPTION:
After ethics committee approval and parental consent were obtained, 119 patients undergoing genitourinary surgery or inguinal hernia repair under general anesthesia, were included in study. Patients with head or neck anomalies, syndromic patients, patients undergoing emergency surgery and patients with a history of difficult airway were excluded from the study. Patients were grouped according to their ages; Group I (1-2 years,n=38), Group II (3-5 years,n=46) and Group III (6-8 years,n=35). USG measurements were performed following sevoflurane induction in groups I and II. In group III, USG measurements were performed following premedication with intravenous midazolam 0.05 mg/kg . Thyrohyoid distance, glottic and subglottic diameters were measured with ultrasonography. The size of the endotracheal tube according to Bae's formula ( internal diameter of Endotracheal tube = 0.705 x subglottic diameter - 0.091) was calculated and recorded. Before intubation, endotracheal tube (cuffed/uncuffed) was selected using age-related formulas. In group II, anaesthesia induction was achieved with propofol 2 mg/kg. In all groups, endotracheal intubation was achieved with fentanyl 2μg/kg and rocuronium 0.6 mg/kg. Endotracheal tube size was considered as optimal when a leak was detected at 20-30cmH₂O inflation pressures. If a resistance was felt in the subglottic region, the tube was exchanged with a smaller and was exchanged with a larger (0.5 mm) size if a leak occurred at inflation pressures lower than 20cmH₂O. Intubation duration , Cormack-Lehane scores and Intubation Difficulty Scale scores were recorded. For comparison of age related formula and Bae 's formula, only patients who were intubated with un-cuffed endotracheal tube were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 1 and 8 years
* Elective surgery

Exclusion Criteria:

* Patients with head or neck abnormalities
* Syndromic patients
* Emergency surgery and patients with a
* History of difficult airway
* Allergy to ultrasound gel

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of difficult intubation (determined with Intubation Difficulty Scale) in patients who have short thyrohyoid distance | three years
Consistency of endotracheal tube sizes selected with aged related formulas and with ultrasonographic measurement of subglotic diameter | three years

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided